CLINICAL TRIAL: NCT04096430
Title: Evaluation of Effectiveness of Child-oriented Goal-setting in Paediatric Rehabilitation (the ENGAGE Approach): A Pragmatic Cluster Randomized Controlled Trial and Economic Analysis
Brief Title: Evaluation of Effectiveness of Child-oriented Goal-setting in Paediatric Rehabilitation (the ENGAGE Approach)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00090963
Record Dates: First submitted 2019-08-14; First posted 2019-09-19 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder; Neurodevelopmental Disorders; Cerebral Palsy
MeSH Terms: conditions — Autism Spectrum Disorder; Neurodevelopmental Disorders; Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: We will use a pragmatic, cluster randomized controlled trial (RCT) design with therapists randomized to one of two groups; the ENGAGE intervention group or the usual care control group.
Who Masked: Outcomes Assessor
Masking Description: Trained assessors, blinded to group allocation, will complete the measures with families. Family members will be blinded to all initial responses on the measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENGAGE approach (child-oriented goal-setting) (Experimental): Therapists will receive training on our principles-based goal setting approach and strategies in the goal setting toolbox. Training will include an overview of tools and strategies including the Perceived Efficacy and Goal Setting Tool (PEGS) and the Pediatric Activity Card Sort (PACS). In addition, we will provide training on Goal Attainment Scaling and administration of the Canadian Occupational Performance Measure (COPM). We will introduce simple strategies to assist children in identifying goals and to ensure ongoing focus on goals using principles of motivational interviewing, strategies to assess and nurture perceived competence (self-efficacy), and child-friendly feedback strategies on goal-related performance.
  Interventions: Behavioral: ENGAGE approach (child-oriented goal-setting)
- Usual care (No Intervention): The control group will comprise of usual care.

INTERVENTIONS:
Behavioral: ENGAGE approach (child-oriented goal-setting) — See description of experimental arm.
  Arms: ENGAGE approach (child-oriented goal-setting)

SUMMARY:
Children with disabilities often access rehabilitation services to improve their abilities to participate in everyday activities. Goal-directed therapy is considered an important therapeutic strategy to achieve outcomes that are meaningful to families. Not a lot is known about the effects of goal setting on rehabilitation outcomes. Strategies to help children participate in the goal-setting process are rarely used in clinical practice. The aim of this project is to test the effects of a child-focussed goal setting approach, Enhancing Child Engagement in Goal Setting (ENGAGE), on therapy outcomes. Service use and the cost vs. benefits of the ENGAGE approach compared to usual practice will also be examined. Children with neurodevelopmental disabilities aged 5-12 years old (n=96) who access paediatric rehabilitation services at six rehabilitation sites will participate. Therapists (n=24) at participating sites in Alberta, Canada will be randomized into 1) the ENGAGE intervention group or 2) the usual therapy practice control group. Children will participate in the ENGAGE approach to goal setting or usual practice based on the allocation of their therapist. This study will determine if the ENGAGE approach to goal setting affects child goal performance, satisfaction with goal performance, functional abilities, participation, and parent and child quality of life. The investigators will also evaluate differences in parent and child quality of life in relation to parent costs (e.g., absenteeism, presenteeism, travel costs) and compare amount of therapy time between the two groups to see which approach is more cost-effective and efficient. After the study, children, parents and therapists will be asked to discuss aspects that influenced effective implementation of the ENGAGE approach. This study could provide evidence to improve meaningful child and family outcomes in paediatric rehabilitation and improve efficiency of paediatric rehabilitation services.

DETAILED DESCRIPTION:
PURPOSE:

This pragmatic trial aims to improve health outcomes for children with neurodevelopmental disabilities (NDD) using a novel therapist-targeted, theory-driven, evidence-based approach to goal setting, the Enhancing Child Engagement in Goal Setting (ENGAGE) approach. This study includes an economic analysis and service utilization component and an implementation process analysis to evaluate cost-effectiveness and to support long-term sustainability.

RESEARCH QUESTIONS:

Primary question: Does ENGAGE improve children's engagement in therapy, goal-related performance (primary outcome), functional abilities, participation in home, school and/or community, and child and caregiver quality of life compared to the current standard of care?

Secondary questions: 1) What goal, child, family and therapist factors mediate and/or moderate the effects of ENGAGE on the above intervention outcomes? and 2) Does ENGAGE improve cost effectiveness from the perspectives of parents and service delivery efficiency compared to the current standard of care?

METHODOLOGY/IMPLEMENTATION STRATEGY AND EVALUATION:

Study design: A pragmatic, cluster randomized controlled trial (RCT) design will be used with therapists randomized to one of two groups; the ENGAGE intervention group or the usual care control group. The RCT will be a six-site trial with two groups (ENGAGE training absent/present) with two periods of post-intervention assessment (immediate post-treatment and 3-month follow-up). The trial will take place within established public paediatric rehabilitation sites in Alberta. An economic analysis consisting of a cost-benefit analysis from the perspectives of parents and a comparison of service utilization costs will be conducted in conjunction with the RCT. To facilitate more widespread implementation, a qualitative process evaluation will be conducted to delineate core versus peripheral components of the intervention, and therapist, child and parent perspectives on the contextual features that influenced implementation.

Sample: The sample size will be 96 children (12 therapists as clusters per group and 4 children per therapist) at six sites. Based on the investigators' pilot work, it is anticipated that child dropout from the pre-post intervention period will be minimal (i.e., less than 5%). A target change score of 2.0, a clinically significant change on the COPM (primary outcome), with a standard deviation of 2.75 corresponds to an effect size of 0.723 for the comparison of means. A sample size of 96 will result in an effect size of at least 0.682 in the primary outcome (COPM performance rating) with alpha=0.05 and 80% power assuming an intra-cluster correlation (ICC) of 0.1 using a two-sided, cluster adjusted, t-test for the comparison of means. An ICC of 0.1 was selected based on results of a previous cluster RCT with children with cerebral palsy (ICCs between 0.08 to 0.13). Since therapist attrition is possible over the duration of the study, the sampling strategy was designed so that a cluster size of 11 would still provide 80% power to detect an effect size of 0.716, below the target effect size. Smaller effect sizes will be detectable if the ICC is smaller than 0.1. The sample size was adjusted from 88 to 96 to allow for an 8% loss to follow-up (1 therapist, 4 children per group). The investigators do not anticipate retention issues for the baseline and post-intervention assessments (primary evaluation period). The probability of loss to follow-up may increase at the 3-month follow-up assessment. The estimate of loss to follow-up is based on the investigators' experience with trials with children with disabilities.

Inclusion criteria are children who 1) are 5-12 years old, 2) are referred to PT and/or OT for a period of direct treatment, and 3) speak English. Further inclusion/Exclusion criteria can be found in the protocol in documents section.

Recruitment: Over 18 months, children (n=96) will be sequentially recruited by 24 therapists from six paediatric Alberta rehabilitation sites (4 children per therapist).

Randomization: A computer-generated, permuted-block randomization sequence using site as a stratification variable will be used to allocate 24 OTs and PTs across 6 sites to the ENGAGE or control group to ensure balanced groups.

Study groups: Intervention Group - Therapists will receive training on our principles-based goal setting approach and strategies in the goal setting toolbox. Control group - The control group will comprise usual care. With the exception of the strategies outlined in ENGAGE, rehabilitation interventions used to achieve identified goals will not vary from usual practice. Consistent with a pragmatic trial, this approach will enable us to evaluate effectiveness of ENGAGE in typical clinical settings. .

Treatment duration and intensity for both groups will differ based on nature of goals, treatment strategies, and family preference. It is anticipated that treatment block lengths will vary from 3-8 sessions over 2-8 weeks, representing typical clinical variation.

Fidelity monitoring- Following the training, the strategies used by ENGAGE therapists will be tracked to evaluate treatment fidelity prior to recruiting participants. Feedback will be provided as needed to therapists as part of the implementation plan to facilitate ongoing and consistent use of the intervention strategies. Treatment frequency, intensity, intervention strategies, and feedback frequency and mechanisms will be documented by therapists at each treatment session. Co-interventions will be monitored for each participant. Recruitment and formalized data collection will begin once intervention therapists at the site achieve an acceptable level of fidelity defined as adherence to ENGAGE principles at least 90% of the time. For example, the extent children are involved in identifying their own goals will be monitored and how often therapists use feedback on goal-related performance at each treatment session. Practices will also be monitored in the control group using an open-ended form to prevent contamination from exposure to ENGAGE principles. Ongoing documentation of practices and monitoring will be used to evaluate the need for additional or different implementation support in the intervention group and to enable comparison of group practices.

During ENGAGE training and throughout the study the investigators will reinforce that intervention therapists need to avoid discussion of principles and practices with the control group therapists. Therapists will complete a questionnaire about their typical practices with respect to goal setting at the beginning of the training session (intervention) and orientation (control). These responses will identify if the control group therapists deviate from their approach to goal setting used at baseline over the course of the study and allow for between group comparisons of strategy use.

Data collection and Outcomes: Identical assessments will be conducted at 1) baseline (pre-treatment), 2) post-treatment (within 10 days), and 3) at 3-months post-treatment.

Primary outcome measure is goal performance, satisfaction with performance, goal attainment (Canadian Occupational Performance Measure (COPM)). All data will be entered into REDCap.

An economic analysis consisting of a cost benefit analysis from the family perspective will be conducted in conjunction with this trial. Costs related to ENGAGE relative to typical care will be tracked using a therapy session questionnaire for both groups. In addition, total costs incurred per child during the intervention will be determined by multiplying therapist direct and indirect (e.g., documentation) time by a corresponding unit price. Mean cost per child will then be calculated for each group. Costs from the family perspective will be tracked using a parent questionnaire and outcomes will be parent and child quality of life measures.

Analysis: Data and demographic characteristics will be described (e.g., means, standard deviations) for both groups. Change scores (post minus pre, follow-up minus post) will be summarized for each outcome, with COPM changes post intervention as the primary analysis (Question 1) and the other outcomes as secondary analyses. For each change score and outcome, a cluster adjusted t-test will be used to compare mean change score between groups (ENGAGE, control). A confidence interval will be reported for the difference between group mean scores. Mixed effects linear regression models on all outcomes will include group and time (fixed effects), a therapist random effect (to adjust for the clustering), and a child random effect (to adjust for repeated measures on each child). Time will be a categorical variable so that post and follow-up times can be compared with pre-treatment assessments. A time by group interaction will also be considered to assess the effects of group.

Question 2: Mixed effects multiple linear regression models similar to the above will also be developed for each outcome with the additional variables of site, site by group as an interaction (to assess site effect) and other theoretically important variables (e.g., cognitive abilities, age, parenting style) as covariates.

Question 3: Mean cost per child and the mean effectiveness result per child for each group will be represented in an incremental cost-effectiveness ratio (ICER) - the ratio of the difference between groups in mean cost per patient to the difference in mean effectiveness using the two quality of life measures (CarerQol and KIDSCREEN) as outcomes. Extensive sensitivity analysis including probabilistic sensitivity analysis will be undertaken to test robustness of the results.

Process evaluation: Semi-structured interviews will be conducted during post-intervention assessment with pairs of parent and child participants (n=24 pairs from the ENGAGE condition; n=12 pairs from the control condition), stratified by centre, child age and child diagnosis to ensure variability in the sample. Therapists (n=24) at each of the six sites will also participate in qualitative interviews to explore their experiences with the ENGAGE approach and the implementation process.The CFIR (Consolidated Framework for Implementation Research) framework will be used in conjunction with the Theoretical Domains Framework to sensitize the researchers to known barriers and facilitators to implementation. Interviews will be audio-recorded, professionally transcribed, and last approximately 45-60 minutes. Data will be analyzed using inductive thematic analysis. Journaling will be used throughout data collection and analysis to record preliminary themes/ideas about the data, experiences in the research process and reasoning around decisions in data collection and analysis, and to facilitate research reflexivity.

ELIGIBILITY:
Inclusion criteria are children with a diagnosed disability who:

1. are between the ages of 5-12 years
2. are able to engage in the goal-setting process (determined by therapists)
3. are referred to PT and/or OT for a period of direct treatment
4. speak English.

Children will be excluded from the trial if:

1. the parent or guardian who attends therapy does not speak English
2. the child has a diagnosis that suggests developmental regression
3. the child has uncontrolled seizures (i.e., seizure within the past 2 months).

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Goal performance and satisfaction will be measured using the Canadian Occupational Performance Measure (COPM). | 1) baseline (pre-treatment), 2) post-treatment (within 10 days of completing therapy), and 3) at 3-months post-treatment
  Change in the COPM will be examined between baseline (pre-treatment) and post-treatment (within 10 days of completing therapy), and post-treatment (within 10 days of completing therapy) and 3-months post-treatment. The COPM is an interview style measure in which a child is asked by an assessor to identify goal areas and then rate their current level on a 1 to 10 scale as far as importance, satisfaction and performance. A higher score represents a more favorable outcome.

SECONDARY OUTCOMES:
Child engagement in therapy will be measured using the Pediatric Rehabilitation Intervention Measure of Engagement (PRIME-SP). | 1) baseline (pre-treatment), 2) post-treatment (within 10 days), and 3) at 3-months post-treatment
  Change in the (PRIME-SP) will be examined between baseline (pre-treatment) and post-treatment (within 10 days of completing therapy), and post-treatment (within 10 days of completing therapy) and 3-months post-treatment.
Perceived confidence will be measured using the Belief in Goal Self-Competence Scale [BiGSS]. | 1) baseline (pre-treatment), 2) post-treatment (within 10 days), and 3) at 3-months post-treatment
  Change in the BIGSS will be examined between baseline (pre-treatment) and post-treatment (within 10 days of completing therapy), and post-treatment (within 10 days of completing therapy) and 3-months post-treatment. BIGSS assess percieved using a 10-point Likert scale ("How confident do you feel that you can do this activity?). A higher score represents a more favorable outcome.
Goal related performance will be measured using the Goal Attainment Scaling (GAS). | 1) baseline (pre-treatment), 2) post-treatment (within 10 days), and 3) at 3-months post-treatment
  Change in GAS will be examined between baseline (pre-treatment) and post-treatment (within 10 days of completing therapy), and post-treatment (within 10 days of completing therapy) and 3-months post-treatment.
Participation for young children will be measured using the Participation and Environment Measure for Children & Youth (PEM-CY). | 1) baseline (pre-treatment), 2) post-treatment (within 10 days), and 3) at 3-months post-treatment
  Change in the PEM-CY will be examined between baseline (pre-treatment) and post-treatment (within 10 days of completing therapy), and post-treatment (within 10 days of completing therapy) and 3-months post-treatment. This questionnaire is completed by a child (if 8 years or older) or parent. The participant responds to whether they have performed the activity in the last few weeks, who they did it with, where they did it and how much they enjoyed it.
Quality of life for children will be measured using the KIDSCREEN-27. | 1) baseline (pre-treatment), 2) post-treatment (within 10 days), and 3) at 3-months post-treatment
  Change in the KIDSCREEN-27 will be examined between baseline (pre-treatment) and post-treatment (within 10 days of completing therapy), and post-treatment (within 10 days of completing therapy) and 3-months post-treatment. The KIDSCREEN-27 contains 27 items covering five dimensions: physical well-being (5 items), psychological well-being (7 items), parent relations and autonomy (7 items), social support and peers (4 items), and school (4 items). Each item rates frequency of behaviours/feelings or intensity of attitudes on a 5-point scale, with a higher score reflecting a more favorable outcome.
Caregiver quality of life will be measured with the Caregiver Quality of Life (CarerQol-7D). | 1) baseline (pre-treatment), 2) post-treatment (within 10 days), and 3) at 3-months post-treatment
  Change in CarerQol-7D will be examined between baseline (pre-treatment) and post-treatment (within 10 days of completing therapy), and post-treatment (within 10 days of completing therapy) and 3-months post-treatment. CarerQol is a 7-item questionnaire that evaluates the subjective burden experienced by caregivers across seven dimensions, including fulfillment, relational problems, mental health, daily activities, financial, physical health and support along with overall well-being on a VAS scale.
Functional abilities will be measured with the Pediatric Evaluation of Disability Inventory (PEDI-CAT). | 1) baseline (pre-treatment), 2) post-treatment (within 10 days), and 3) at 3-months post-treatment
  Change in the PEDI-CAT will be examined between between baseline (pre-treatment) and post-treatment (within 10 days of completing therapy), and post-treatment (within 10 days of completing therapy) and 3-months post-treatment. The PEDI-CA T includes domains that align with the I CF-CY domains of activity (daily activities, mobility, social/cognitive) and participation. A parent of each participant will complete the content-balanced version of the PEDI-CA T using iPads at each site. An algorism based on item response theory selects items to minimizes the number ofresponses required, so parents answer up to -30 items/domain.

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Pritchard-Wiart, PhD, Principal Investigator — University of Alberta, Faculty of Rehabilitation Medicine
Locations (6):
- Canada (6):
  - Renfrew Educational Services, Calgary, Alberta
  - Society for Treatment of Autism, Calgary, Alberta
  - Children's Rehabilitation Services, Alberta Health Services, Camrose, Alberta
  - Centre for Autism Services Alberta, Edmonton, Alberta
  - Children's Rehabilitation Services, Alberta Health Services, Grande Prairie, Alberta
  - Children's Rehabilitation Services, Alberta Health Services, Red Deer, Alberta

IPD SHARING:
Plan to Share IPD: No